CLINICAL TRIAL: NCT01985217
Title: Prevalence of Digestive Carriage of Integrons to Resistance in Two Populations in Limousin
Brief Title: Prevalence of Digestive Carriage of Integrons
Acronym: APIHA
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I07020
Record Dates: First submitted 2013-11-04; First posted 2013-11-15 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Bacterial Resistance to Antimicrobial

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Bacterial resistance to antimicrobials is an increasing problem. Doctors occasionally face genuine therapeutic dead-ends, when attempting to cure nosocomial infections and, more and more frequently, community-acquired infections. Mastering antimicrobial resistance diffusion is nowadays a major Public Health issue.

DETAILED DESCRIPTION:
Struggling against bacterial resistance to antimicrobials lays on three main measures:

* individual and collective hygiene.
* proper antibiotics practices, which could help reduce antibiotic selective pressure.
* better understanding of bacterial resistance mechanisms and resistance gene transfer between bacteria.

Integrons, gene capture and expression systems, are recognised as major players in resistance gene transfer, which accounts for the greater part of resistance emergence and dissemination. Integrons are typically described in Gram negative bacteria, isolated in man, environmental settings and animals. They encode resistances to nearly every class of antimicrobials. A strong link between integrons and resistance to multiple antibiotic compounds has been described and integron detection is a relevant indicator of resistance to multiple antibiotics.

The investigators project offers to study the impact of antibiotics on the frequency of integron intestinal carriage in the Limousin region and the genetic communities between the two groups.

This study will use an innovative real-time PCR technique to detect integrons directly in the sample without using traditional culture-based techniques. The investigators hope to detect new integron-carriers, notably patients for whom integrons are borne by non or poorly cultivable bacteria. Stool samples will be taken from two groups of subjects : 246 intensive-care unit patients under high antibiotic selective pressure, compared with 246 healthy individuals representative of the community, under a more usual selective pressure. In both groups, antibiotic consumption will be fully documented.

ELIGIBILITY:
Inclusion Criteria:

* adults > 18 years
* patients Hospitalized in intensive care unit for at least 48 hours, including one antibiotic was found at least in the background (<3 months).
* patients followed by the Department for Work and Health for bacteriological examination of stool
* possible information about antibiotic therapy provided

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: people working in the hospital kitchen
Sampling Method: Non-Probability Sample
Enrollment: 492 (Actual)
Dates: Start 2009-08; Primary Completion 2012-04 (Actual); Study Completion 2013-12

PRIMARY OUTCOMES:
Positive PCR | day 1
  * From the "conventional", a subject is found integrons carrying resistance when the PCR is positive on at least one bacterial strain previously isolated.
  * According to the "direct" approach, a subject is considered integrons carrying resistance when the PCR is positive in the DNA extracted directly from feces or broth enrichment.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Virologie, Limoges, France